CLINICAL TRIAL: NCT02045849
Title: A Single-Center, Three-Part, Open Label Study to Evaluate the Relative Bioavailability of Two Formulations, Food Effect, and Interaction With Itraconazole Following Single Dose of GSK2140944 in Healthy Subjects and Effect of Food on Safety, Tolerability, and Pharmacokinetics Following Multiple Doses of GSK2140944 in Healthy Elderly Subjects
Brief Title: Relative Bioavailability, Safety, Tolerability, Pharmacokinetics (PK) and Food Effect Study of GSK2140944 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 117349
Record Dates: First submitted 2014-01-23; First posted 2014-01-27 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Infections, Bacterial
Keywords: pharmacokinetics; GSK2140944; tolerability; drug interaction; safety; itraconazole; elderly healthy subjects; food effect; relative bioavailability
MeSH Terms: conditions — Bacterial Infections | interventions — gepotidacin; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part 1 (Experimental): Subjects will receive either GSK2140944 1500 mg (500 mg x 3) capsules under fasted conditions or GSK2140944 1500 mg (750 mg x 2) tablets under fasted conditions or GSK2140944 1500 mg (750 mg x 2) tablets under fed conditions as per the randomization schedule in each of the three periods with a washout period of at least 3 days between the doses. There will also be a follow-up visit within 5-7 days after the last dose of study drug.
  Interventions: Drug: GSK2140944 capsule; Drug: GSK2140944 tablet
- Part 2 (Experimental): Subjects will receive a single dose of GSK2140944 1500 mg (tablet or capsule) on Day 1 followed by a repeat dose of Itraconazole 200 mg once daily for 6 days from Day 4 to Day 9. On Day 7, subjects will receive a single dose of GSK2140944 1500 mg (tablet or capsule) one hour after the dose of Itraconazole. There will also be a follow-up visit within 5-7 days after the last dose of study drug.
  Interventions: Drug: GSK2140944 capsule; Drug: GSK2140944 tablet; Drug: Itraconazole capsule
- Part 3 (Experimental): Subjects in Group 1 will receive GSK2140944 1500 mg (750 mg x 2) tablets twice daily from Day 1 to Day 5 under fasting and fed conditions in Period I and Period II, respectively. Subjects in Group 2 will receive GSK2140944 1500 mg (750 mg x 2) tablets twice daily from Day 1 to Day 5 under fed and fasting conditions in Period I and Period II, respectively. There will be a washout of at least 7 days between the periods. Subjects will have a follow up visit 5-7 days after the last dose of study drug in both the groups.
  Interventions: Drug: GSK2140944 tablet

INTERVENTIONS:
Drug: GSK2140944 capsule — Immediate release capsule containing GSK2140944 and inactive formulation excipients with a unit dose strength of 500 mg
  Arms: Part 1; Part 2
Drug: GSK2140944 tablet — Immediate release tablet containing GSK2140944 and inactive formulation excipients with a unit dose strength of 750 mg
Drug: Itraconazole capsule — Capsule containing Itraconazole with a unit dose strength of 100 mg
  Arms: Part 2

SUMMARY:
This study will be conducted in three parts (Part 1, Part 2 and Part 3). Part 1 of this study will evaluate the relative bioavailability of a single dose of GSK2140944 tablet formulation compared to the reference capsule formulation under fasted conditions. The effect of food on the pharmacokinetics (PK) of a single dose of the tablet formulation will also be assessed. Part 2 will evaluate the effect of repeat doses of itraconazole on the pharmacokinetics of GSK2140944 following a single dose. A decision will be made whether to use the current capsule formulation or the new tablet formulation in Part 2 based upon the safety and PK data obtained from Part 1. Part 3 is conditionally based upon progression of the tablet formulation from Part 1 and will evaluate the effect of food on the safety, tolerability, and pharmacokinetics of the tablet formulation following multiple doses in elderly healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator feels and documents that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Part 1 and 2: Male or female between 18 and 64 years of age inclusive, at the time of signing the informed consent. Part 3: Male or female subjects at least 65 years of age or older at the time of signing the informed consent.
* A female subject is eligible to participate if she is of: non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea. To confirm post-menopausal status, a blood sample for simultaneous follicle stimulating hormone (FSH) >40 milli-International Units (MIU)/milliliter (mL) and estradiol <40 picograms (pg)/mL (<147 picomoles [pmol]/liter [L]) is confirmatory. Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods. This criterion must be followed from the time of the first dose of study medication until the final follow-up visit.
* Body weight >=50 kilograms (kg) and body mass index (BMI) within the range 19 - 31 kg/meter square (m^2) (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Alanine amino transferase (ALT), alkaline phosphatase and bilirubin <=1.5xUpper Limit of Normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).

Exclusion Criteria:

Criteria Based Upon Medical Histories

* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Any clinically significant central nervous system (e.g., seizures), cardiac, pulmonary, metabolic, renal, hepatic or gastrointestinal conditions or history of such conditions that, in the opinion of the investigator may place the subject at an unacceptable risk as a participant in this trial or may interfere with the absorption, distribution, metabolism or excretion of drugs.
* History of photosensitivity to quinolones.
* Use of systemic antibiotic within 30 days of screening
* Previous exposure to GSK2140944
* Confirmed history of C-difficile diarrhea.
* History of tendon rupture.
* History of drug abuse within 6 months of the study.
* History of smoking or use of nicotine containing products within 3 months of screening, or a positive urine cotinine indicative of smoking at screening.
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 grams of alcohol: 12 ounces (360 mL) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* History of sensitivity to heparin or heparin-induced thrombocytopenia (if the clinical research unit uses heparin to maintain intravenous cannula patency).

Criteria Based Upon Diagnostic Assessments

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening or positive Human Immunodeficiency Virus (HIV) antibody.
* A screening or Day -1 urinalysis positive for protein or glucose (greater than 1+ findings of protein or glucose).
* A serum creatinine value that is increased by more than 0.2 milligram (mg)/deciliter (dL) (or 15.25 micromoles/L) between screening and Day -1.
* For Part 3 Only: Neutrophil count <2000 cells/microliter (a single repeat is allowed for eligibility determination).
* A positive urine test for drugs of abuse or alcohol (or alcohol breath test) at screening or at Day -1.
* Exclusion criteria for screening and baseline ECG (a single repeat is allowed for eligibility determination) as follows: Heart rate: <40 and >100 beats per minute (bpm) for males and <50 and >100 bpm for females; PR Interval: <120 and >220 milliseconds (msec); QRS duration: <70 and >100 msec; QT duration corrected for heart rate by Bazett's formula (QTcB) or QT duration corrected for heart rate by Fridericia's formula (QTcF) interval>450 msec. Evidence of previous myocardial infarction (does not include ST segment changes associated with repolarization). Any conduction abnormality (including but not specific to left or right complete bundle branch block, atrioventricular (AV) block [2nd degree or higher], Wolf Parkinson White [WPW] syndrome), sinus pauses> 3 seconds, non-sustained or sustained ventricular tachycardia (>=3 consecutive ventricular ectopic beats) or any significant arrhythmia which, in the opinion of the principal investigator and GSK medical monitor, will interfere with the safety of the individual subject.

Other Criteria

* Donation of blood in excess of 500 mL within 12 weeks prior to dosing or participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Unwillingness to commit to avoid excessive exposure to sunlight (or exposure to a tanning bed) which would cause a sunburn reaction from first dose up to and including the follow-up visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2014-01-28 (Actual); Primary Completion 2014-08-21 (Actual); Study Completion 2014-08-21 (Actual)

PRIMARY OUTCOMES:
Part 1: Composite of PK parameters following GSK2140944 administration in fasted and fed state | Day 1 (Pre-dose, 0.25h, 0.5h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 12h, 24h, 36h, and at 48h)
  PK parameters will include area under the concentration-time curve (AUC) from time zero (pre-dose) extrapolated to infinite time AUC(0-infinity), AUC from time zero to last quantifiable concentration AUC(0-t), relative bioavailability of drug (Frel), maximum observed concentration (Cmax), time of occurrence of Cmax (tmax), lag time before observation of drug concentration (tlag) and terminal phase half-life (t1/2) in the fasted state; AUC(0-infinity), AUC(0-t), tmax, tlag and Cmax after moderate fat meal.
Part 2: Composite of PK parameters of GSK2140944 following repeat oral dosing of itraconazole | Day 1 and Day 7 (Predose, 0.25h, 0.5h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 12h, 24h, 36h, and 48h post dose and also at 60h and 72h post dose on Day 7
  PK parameters will include AUC(0-infinity), AUC(0-t), tmax, tlag and Cmax of GSK2140944.
Part 3: Safety and tolerability of GSK2140944 as assessed by adverse events (AEs) | Approximately 8 weeks
Part 3: Safety and tolerability of GSK2140944 as assessed by review of concomitant medications | Approximately 8 weeks
Part 3: Safety and tolerability of GSK2140944 by laboratory assessments | Approximately 8 weeks
  Laboratory assessments will include hematology, clinical chemistry, urinalysis parameters
Part 3: Safety and tolerability of GSK2140944 as assessed by 12-lead electrocardiograms (ECGs) | Approximately 8 weeks
  All 12-lead ECGs will be obtained after the subject has rested in a supine position for at least 10 minutes
Part 3: Safety and tolerability of GSK2140944 as assessed by vital signs | Approximately 8 weeks
  Vital signs will be measured for subjects in supine position and will include systolic and diastolic blood pressure, pulse rate and temperature

SECONDARY OUTCOMES:
Part 1: Safety and tolerability of GSK2140944 as assessed by AEs | Approximately 7 weeks
Part 1: Safety and tolerability of GSK2140944 as assessed by review of concomitant medications | Approximately 7 weeks
Part 1: Safety and tolerability of GSK2140944 by laboratory assessments | Approximately 7 weeks
  Laboratory assessments will include hematology, clinical chemistry, urinalysis parameters
Part 1: Safety and tolerability of GSK2140944 as assessed by 12-lead ECGs | Approximately 7 weeks
  All 12-lead ECGs will be obtained after the subject has rested in a supine position for at least 10 minutes
Part 1: Safety and tolerability of GSK2140944 as assessed by vital signs | Approximately 7 weeks
  Vital signs will be measured for subjects in supine position and will include systolic and diastolic blood pressure, pulse rate and temperature
Part 2: Safety and tolerability of GSK2140944 as assessed by AEs | Approximately 6 weeks
Part 2: Safety and tolerability of GSK2140944 by laboratory assessments | Approximately 6 weeks
  Laboratory assessments will include hematology, clinical chemistry, urinalysis parameters
Part 2: Safety and tolerability of GSK2140944 as assessed by 12-lead ECGs | Approximately 6 weeks
  All 12-lead ECGs will be obtained after the subject has rested in a supine position for at least 10 minutes
Part 2: Safety and tolerability of GSK2140944 as assessed by vital signs | Approximately 6 weeks
  Vital signs will be measured for subjects in supine position and will include systolic and diastolic blood pressure, pulse rate and temperature
Part 3: Composite of PK parameters of GSK2140944 following repeat oral dosing of GSK2140944 | Day 3 and Day 4 (Pre-dose), Day 5 (Predose, 0.25h, 0.5h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 12h, 24h, 36h, and at 48h)
  PK parameters will include AUC over the dosing interval (0-tau), tmax, tlag, t1/2, pre-dose (trough) concentration at the end of the dosing interval (Ctau) and Cmax of GSK2140944

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Tiffany C, Dumont EF, Hossain M, Srinivasan M, Swift B. Pharmacokinetics, safety, and tolerability of gepotidacin administered as single or repeat ascending doses, in healthy adults and elderly subjects. Clin Transl Sci. 2022 Sep;15(9):2251-2264. doi: 10.1111/cts.13359. Epub 2022 Jul 13. PMID 35769034
- See also: Results for study 117349 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/117349?search=study&study_ids=117349#rs
- Available data/document: Informed Consent Form: 117349 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 117349 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 117349 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 117349 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 117349 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 117349 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 117349 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register